CLINICAL TRIAL: NCT05095779
Title: Monetary Incentives to Promote Engagement With the Oklahoma Tobacco Helpline in Counties Experiencing Persistent Poverty
Brief Title: Incentives for Oklahoma Tobacco Helpline Engagement in Persistent Poverty Counties
Acronym: CLIMB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Tobacco Settlement Endowment Trust (TSET) (Unknown); National Cancer Institute (NCI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13859; P30CA225520 (NIH); K01MD015295 (NIH); R25MD011564 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Cigarette Smoking; Nicotine Dependence
Keywords: Persistent Poverty; Smoking Cessation; Financial Incentives; Contingency Management; Tobacco Helpline; Tobacco Quitline; Socioeconomic Status
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oklahoma Tobacco Helpline (OTH) (Active Comparator): Participants randomized to OTH will be offered coaching calls and nicotine replacement therapy.
  Interventions: Behavioral: Coaching calls; Drug: Nicotine replacement therapy
- OTH + Financial Incentives (OTH+FI) (Experimental): Participants will receive standard OTH care (coaching calls + nicotine replacement therapy) and escalating financial incentives for completing up to 5 coaching calls.
  Interventions: Behavioral: Coaching calls; Drug: Nicotine replacement therapy; Behavioral: Financial Incentives

INTERVENTIONS:
Behavioral: Coaching calls — OTH coaching calls
Drug: Nicotine replacement therapy — 8 weeks of nicotine replacement therapy
Behavioral: Financial Incentives — Escalating financial incentives for completing up to 5 coaching calls
  Arms: OTH + Financial Incentives (OTH+FI)

SUMMARY:
The proposed pilot project is designed to evaluate the feasibility and potential efficacy of offering small financial incentives for the completion of smoking cessation counseling and self-reported abstinence at follow-up among Oklahoma Tobacco Helpline (OTH) callers living in persistent poverty counties (PPCs). The study will enroll at least 160 adults who reside in any of the 16 persistent poverty counties in Oklahoma, who are seeking smoking cessation treatment through the OTH.

DETAILED DESCRIPTION:
The proposed randomized controlled trial will enroll adults who are seeking smoking cessation treatment through the OTH and who reside in any of the 16 PPCs in Oklahoma. Participants will be randomly assigned to OTH (coaching calls + nicotine replacement therapy) or OTH plus escalating financial incentives (OTH+FI) for completing up to 5 counseling calls over 8 weeks. Feasibility outcomes for the incentives-based intervention will focus on counseling call completions, follow-up assessment completion, smoking cessation, and incentive costs. Potential effectiveness will be evaluated based on comparisons of counseling call completions over the first 8 weeks post-enrollment and rates of self-reported smoking abstinence through 12 weeks post-enrollment (4 weeks after incentives have ended) in OTH+FI relative to OTH alone.

ELIGIBILITY:
Inclusion Criteria:

1. Contact the OTH seeking smoking cessation treatment
2. Reside in any of the 16 PPCs in Oklahoma (Adair, Caddo, Cherokee, Choctaw, Greer, Harmon, Haskell, Hughes, Johnston, McCurtain, Okfuskee, Payne, Pushmataha, Seminole, Sequoyah, Tillman)
3. Report smoking ≥ 5 cigarettes per day
4. Are ≥ 18 years of age
5. Are able to provide a copy/photo of their ID/driver's license or other documentation of identity and residence
6. Be able to read, speak, and understand English
7. Have no contradictions for NRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darla E. Kendzor, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to investigators upon request, after publication of the primary study findings, and with a data-sharing agreement that specifies the investigator(s) will 1) use the data only for research purposes and not to identify any individual participant, 2) store the data on a secure device (e.g., encrypted, password-protected), and 3) destroy or return the data after completion of the analyses.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be made available to investigators upon request after publication of the primary study findings.
Access Criteria: Data sharing agreement

REFERENCES:
- [Result] Kendzor DE, Davie M, Chen M, Hart J, Frank-Pearce SG, Doescher MP, Alexander AC, Businelle MS, Ogunsanya ME, Sifat MS, Boozary LK. Incentivizing Tobacco Helpline Engagement in Persistent Poverty Counties: A Randomized Trial. Am J Prev Med. 2025 Feb;68(2):336-347. doi: 10.1016/j.amepre.2024.10.014. Epub 2024 Oct 29. PMID 39477130

RESULTS

PARTICIPANT FLOW:
Groups:
- Oklahoma Tobacco Helpline (OTH): Participants randomized to OTH were be offered 5-7 counseling calls and 8 weeks of nicotine replacement therapy.
- Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI): Participants randomized to OTH+FI were offered 5-7 counseling calls and 8 weeks of nicotine replacement therapy. In addition, participants had the opportunity to earn incentives for the completion of up to five OTH coaching calls over the first eight weeks post-enrollment.
Period: Overall Study
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Started | 81 | 84
Completed | 65 | 73
Not Completed | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Oklahoma Tobacco Helpline (OTH): Participants were offered coaching calls and 8 weeks of nicotine replacement therapy.
- Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI): Participants were offered coaching calls and 8 weeks of nicotine replacement therapy. In addition, participants had the opportunity to earn incentives for the completion of up to 5 coaching calls over the first 8 weeks post-enrollment.
- Total: Total of all reporting groups
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI) | Total
Number analyzed (Participants) | 81 | 84 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.49 (13.84) | 46.14 (13.65) | 47.79 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 105
  Male | 29 | 31 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 78 | 80 | 158
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 12 | 20
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 63 | 67 | 130
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81 | 84 | 165
Cigarettes Smoked Per Day (pre-quit) [Mean (Standard Deviation); unit: Cigarettes per day] | 21.41 (11.40) | 20.64 (11.97) | 21.01 (11.67)

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Point Prevalence Abstinence
Description: Self-reported smoking abstinence 7-day point prevalence at 12 weeks post-enrollment (missing considered smoking).
Time Frame: 12 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Oklahoma Tobacco Helpline (OTH): Participants were offered 5-7 coaching calls and 8 weeks of nicotine replacement therapy.
- Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI): Participants were offered 5-7 coaching calls and 8 weeks of nicotine replacement therapy. In addition, participants had the opportunity to earn incentives for the completion of up to 5 coaching calls over the first 8 weeks post-enrollment.
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Number analyzed (Participants) | 81 | 84
Participants | 30 | 44

2. Secondary Outcome: 7-Day Point Prevalence Abstinence
Description: Self-reported 7-day point prevalence abstinence at 8 weeks post-enrollment (missing considered smoking)
Time Frame: 8 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Number analyzed (Participants) | 81 | 84
Participants | 26 | 42

3. Secondary Outcome: Coaching Calls Completed (Total Number)
Description: The total number of coaching calls completed.
Time Frame: First 8 weeks post-enrollment
Measure: Median (Inter-Quartile Range); unit: calls completed
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Number analyzed (Participants) | 81 | 84
calls completed | 2 [1 to 3] | 3 [1 to 4]

4. Secondary Outcome: Completed >=3 Coaching Calls
Description: The proportion of participants who completed at least 3 coaching calls
Time Frame: First 8 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Number analyzed (Participants) | 81 | 84
Participants | 22 | 46

5. Secondary Outcome: Retention
Description: The number of participants who completed the follow-up assessment.
Time Frame: 8 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Number analyzed (Participants) | 81 | 84
Participants | 69 | 71

6. Secondary Outcome: Retention
Description: The number of participants who completed the follow-up assessment.
Time Frame: 12 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Number analyzed (Participants) | 81 | 84
Participants | 65 | 73

7. Secondary Outcome: Incentives Earned
Description: The mean amount of call-contingent incentives earned among participants assigned to the OTH+FI group.
Time Frame: First 8 weeks post-enrollment
Population: Participants in the OTH group did not earn call-contingent incentives.
Measure: Mean (Standard Error); unit: dollars
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
Number analyzed (Participants) | 0 | 84
dollars |  | 60.71 (39.77)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Oklahoma Tobacco Helpline (OTH) | Oklahoma Tobacco Helpline + Financial Incentives (OTH+FI)
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/84
Other Adverse Events (participants affected / at risk) | 0/81 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT05095779/Prot_SAP_000.pdf